CLINICAL TRIAL: NCT06568913
Title: The Outcome of the Thrombopoietin Receptor Agonists in Pediatric Patient With Persistent or Chronic ITP Unresonsive to Steroids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shimaa Abdelhameed Mohamed, Resident of pediatric and neonatology department, Sohag University Hospitals, Sohag University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Soh-Med-24-07-12MS
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Persistent or Chronic ITP Not Respnding to Steroids
Keywords: CBC

STUDY DESIGN:
Intervention Model Description: follow up of platelets count and The outcome of the thrombopoietin receptor agonists in pediatric patient with persistent or chronic ITP unresponsive to steroids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persistent or chronic ITP not responsive to steroids (Experimental): The Outcome of the Thrombopoietin Receptor Agonists in Pediatric Patient With Persistent or Chronic ITP Unresonsive to Steroids
  Interventions: Diagnostic Test: CBC

INTERVENTIONS:
Diagnostic Test: CBC — Platelets counts in pediatric patient with perisistent or chronicITP unresponsive to steroids

SUMMARY:
Immune thrombocytopenic purpura (ITP) is an autoimmune disease characterized by a low platelet count, purpura, and hemorrhagic episodes caused by antiplatelet autoantibodies. The diagnosis is typically made by excluding the known causes of thrombocytopenia. IgG autoantibodies sensitize the circulating platelets. It leads to the accelerated removal of these cells by antigen-presenting cells (macrophages) of the spleen and sometimes the liver or other components of the monocyte-macrophage system. The bone marrow compensates for platelet destruction by increasing platelet production. ITP most often occurs in healthy children and young adults within a few weeks following a viral infection .

New treatment guidelines have supported a shift from corticosteroids and splenectomy to newer medical treatments that mitigate the thrombocytopenia and avoid splenectomy. The thrombopoietin receptor agonists (TPO-RA), romiplostim, eltrombopag have markedly altered the treatment of ITP.

The thrombopoietin receptor agonists (TPO-Ras) romiplostim and eltrombopag have shown high therapeutic activity In primary ITP.

Romiplostim, a thrombopoiesis-stimulating peptibody, represents a new therapeutic option in adult refractory chronic immune thrombocytopenia (ITP). This study aimed to assess the short-term efficacy and safety of romiplostim in children withChronic ITP.

The most commonly reported drug-related adverse effects include headache, nausea, and hepatobiliary laboratory abnormalities. Long-term safety data in children are limited, and studies in adults have not revealed a clinically significant increased incidence of thrombosis, marrow fibrosis, or cataract formation.

TPO-RA do not need to be continued forever; about a third of patients In the first year and about another third after two years have a remission. Whether TPO-RA affect the ITP pathophysiology and directly cause remission remains unclear. This review provides a personal overview of the diagnosis and treatment of ITP with a focus on the mechanism of action of TPO-RA, their place in the treatment algorithm, unique aspects of their clinical use, adverse effects.

ELIGIBILITY:
Inclusion Criteria:

pediatric patients with persistent or chronic Itp on thrombopoietin receptor agonists unresponsive to steroid.

Exclusion Criteria:

Any patient with other causes of thrombocytopenia. Any patient with chronic disease . Any patient with Acute ITP . Any newly diagnosed patient with ITP.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-07-14 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Platelets counts in Pediatric Patient With Persistent or Chronic ITP Unresonsive to Steroids on thrombopoietin receptor agonists | 12 months
  The Outcome of the Thrombopoietin Receptor Agonists in Pediatric Patient With Persistent or Chronic ITP Unresonsive to Steroids

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zaja F, Barcellini W, Cantoni S, Carpenedo M, Caparrotti G, Carrai V, Di Renzo N, Santoro C, Di Nicola M, Veneri D, Simonetti F, Liberati AM, Ferla V, Paoloni F, Crea E, Volpetti S, Tuniz E, Fanin R. Thrombopoietin receptor agonists for preparing adult patients with immune thrombocytopenia to splenectomy: results of a retrospective, observational GIMEMA study. Am J Hematol. 2016 May;91(5):E293-5. doi: 10.1002/ajh.24341. Epub 2016 Apr 4. PMID 26910388
- [Background] Mokhtar GM, Tantawy AA, El Sherif NH. Romiplostim therapy in children with unresponsive chronic immune thrombocytopenia. Platelets. 2012;23(4):264-73. doi: 10.3109/09537104.2011.619601. Epub 2012 Apr 3. PMID 22471399
- [Background] Bussel JB, Soff G, Balduzzi A, Cooper N, Lawrence T, Semple JW. A Review of Romiplostim Mechanism of Action and Clinical Applicability. Drug Des Devel Ther. 2021 May 26;15:2243-2268. doi: 10.2147/DDDT.S299591. eCollection 2021. PMID 34079225
- [Background] Giordano P, Lassandro G, Barone A, Cesaro S, Fotzi I, Giona F, Ladogana S, Miano M, Marzollo A, Nardi M, Notarangelo LD, Pession A, Ruggiero A, Russo G, Saracco P, Spinelli M, Tolva A, Tornesello A, Palladino V, Del Vecchio GC. Use of Eltrombopag in Children With Chronic Immune Thrombocytopenia (ITP): A Real Life Retrospective Multicenter Experience of the Italian Association of Pediatric Hematology and Oncology (AIEOP). Front Med (Lausanne). 2020 Feb 28;7:66. doi: 10.3389/fmed.2020.00066. eCollection 2020. PMID 32181255